CLINICAL TRIAL: NCT05897489
Title: SGLT2 Inhibitors in Adult Patients With Heart Failure Related to Congenital Heart Disease
Brief Title: SGLT2 for Heart Failure in CHD Patients
Acronym: GACH
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23Cardio01
Record Dates: First submitted 2023-05-26; First posted 2023-06-09 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure (HF) in adult patients with congenital heart disease is a major cause of morbidity and mortality. Approximately 30% of patients with significant congenital heart disease will develop signs of heart failure. Heart failure leads to hospitalization and disability with a longer hospital stay and higher health care costs as compared to heart failure patients without congenital heart disease. One-third of deaths in patients with congenital heart disease are attributable to heart failure.

In patients with heart failure and reduced ejection fraction (EF), 2021 ESC recommendations suggest the use of sodium-glucose co-transporter 2 inhibitors (SGLT2i) (dapaglifozin and empaglifozin), a new therapeutic class for heart failure (HF), in a class IA recommendation. In addition to reduced EF, these molecules have shown efficacy in preserved EF, leading to their reimbursement in both preserved and reduced ejection fraction in France.

Unfortunately, given the relatively low number of HF-congenital heart disease, patients, they were not included in previous studies. However, the seriousness of their condition and the absence of therapeutic explain the prescription of SGLT2i in those patients and the likelihood of increased use in the future. This especially underlines the need for safety data in this real-world population.

To date, no data on the safety or efficacy of SGLT2i in HF-congenital heart disease have been published. The results of this study would provide reassurance about the safety of SGLT2i in adult congenital patients and potentially expand the indication of SGLT2i in HF related to congenital heart disease

The objective of this study is to assess on real-life data, through a multicenter registry:

* The efficacy of SGLT2i in patients with heart failure related to congenital heart disease - The indications of SGLT2i use (type of congenital heart disease)
* The safety of SGLT2i (collection of adverse events)

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Congenital heart disease (repaired, unrepaired, or palliated) with clinical heart failure NYHA class II, III, or IV at the time of SGLT2i initiation B59
* Patient in whom SGLT2i therapy has been started within the previous 12 months or is started at the time of the visit.
* Registered to the French social security system

Exclusion Criteria:

* Opposition of the patient to the use of his/her data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with heart failure and congenital heart disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
To evaluate, on real-life data, the efficacy of iSGLT2 in patients with heart failure related to congenital heart disease as defined by improvement in NYHA class and/or change in NT-proBNP. | 6 to 12 months after SGLT2i introduction
  Efficacy of SGLT2i therapy will be assessed by a composite endpoint including NT-proBNP and NYHA class. Thus, a patient with any improvement (decrease) in the biomarker (NT-proBNP) and/or improvement in at least 1 NYHA class will be defined as successful with SGLT2i therapy. The success rate in the target population will be calculated at the end of the study follow-up

SECONDARY OUTCOMES:
To describe the population of adults with congenital heart disease on SGLT2i prescription | 6-12 months after SGLT2i introduction
  The study population will be described by the history of the disease in particular duration of the evolution of the CI
To compare the evolution of biological stress test parameters of SGLT2i in patients with heart failure related to congenital heart disease treated with iSGLT2. | 6-12 months after SGLT2i introduction
  The evolution of the following efficacy parameters between baseline and M6/M12 will be studied : biological parameters (Plasma creatinine at T0 and 6-12 months, Kalemia at T0 and 6-12 months)
Incidence of Treatment-Emergent Adverse Event in patients with heart failure related to congenital heart disease.[Safety and Tolerability] | 6-12 months after SGLT2i introduction
  Tolerance will be studied through the collection of the following adverse events:
  arterial hypotension (BP will be recorded at M0, M6 and M12), hyperkalemia, acute renal failure, recurrent urinary tract infections, ketoacidosis (Discontinuation of treatment for AEs, Cardiovascular hospitalization during the study period, Cardiac transplantation or ventricular assist during the study period)
To evaluate the overall survival of heart failure related to congenital heart disease patients on SGLT2i after 12 months | 6-12 months after SGLT2i introduction
  Overall survival will be assessed at 6 months and 12 months after initiation of treatment. Survival time will be defined as the time in months from initiation of glifozine to death from any cause. Patients who discontinue follow-up before the end of the study follow-up period will be censored at the time of last report.

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No